CLINICAL TRIAL: NCT01742208
Title: A Phase 2, Multicenter, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of LX4211 in Patients With Inadequately Controlled Type 1 Diabetes Mellitus
Brief Title: Safety and Efficacy of Sotagliflozin (LX4211) in Patients With Inadequately Controlled Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-203-T1DM; LX4211.203 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2012-11-20; First posted 2012-12-05 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Sotagliflozin 400 mg - Pioneer Group (Experimental): Sotagliflozin 400 milligram (mg) (two 200 mg tablets), once daily, orally, before breakfast for 29 days; open label administration.
  Interventions: Drug: Sotagliflozin
- Placebo - Expansion Group (Placebo Comparator): Two placebo-matching sotagliflozin tablets, once daily, orally, before breakfast for 29 days; double-blind administration.
  Interventions: Drug: Placebo
- Sotagliflozin 400 mg - Expansion Group (Experimental): Sotagliflozin 400 mg (two 200 mg tablets), once daily, orally, before breakfast for 29 days; double-blind administration.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Participants received sotagliflozin once daily for 29 days. Pioneer Group participants were to have completed dosing prior to any study drug administration in Expansion Groups.
  Other Names: LX4211
  Arms: Sotagliflozin 400 mg - Pioneer Group
Drug: Placebo — Participants received placebo-matching sotagliflozin tablets once daily for 29 days.
  Arms: Placebo - Expansion Group
Drug: Sotagliflozin — Participants received sotagliflozin once daily for 29 days; pioneer participants completed dosing prior to dosing any other study participants.
  Other Names: LX4211
  Arms: Sotagliflozin 400 mg - Expansion Group

SUMMARY:
This Phase 2 study was intended to assess the pharmacodynamics (PD), pharmacokinetics (PK), safety and efficacy of sotagliflozin following daily oral administration for 29 days in participants with type 1 diabetes mellitus (T1DM).

ELIGIBILITY:
Inclusion Criteria:

* Adults >=18 to <=55 years of age
* Confirmed diagnosis of T1DM, diagnosed prior to age 40 years, and for at least 6 months prior to Screening
* Willing to refrain from using carbohydrate counting to adjust insulin during the study
* Willing and able to wear and operate a continuous glucose monitor
* Willing and able to self-assess blood glucose
* Willing and able to provide written informed consent.

Exclusion Criteria:

* History of type 2 diabetes mellitus or diabetes resulting from acromegaly, Cushing's disease, chronic pancreatitis, or pancreatectomy
* Two or more severe episodes of hypoglycemia that required emergency treatment within 3 months prior to Screening
* Use of premixed insulin
* History of diabetic ketoacidosis within 1 year of screening
* Presence of active hepatic disease or clinically significant abnormal liver function tests
* History of chronic pancreatitis
* Participants with a history of heart attack, severe/unstable angina, or coronary revascularization procedure
* History of clinically significant cardiac arrhythmias within 1 year prior to screening
* Participants with congestive heart failure
* Participants with uncontrolled Stage III hypertension
* History of human immunodeficiency virus (HIV) or hepatitis C
* History of illicit drug or alcohol abuse within 12 months prior to Screening
* Use of any investigational agent or device within 30 days prior to Screening or any therapeutic protein or antibody within 90 days prior to Screening
* Use of medication or herbal supplements taken for weight loss within 2 weeks of screening
* Chronic use of any antidiabetic therapy other than insulin within 2 months prior to Screening
* Use of systemic or inhaled corticosteroids within 2 weeks prior to Screening
* Participants who underwent major surgery within 6 months prior to Screening
* Inability or difficulty swallowing whole tablets or capsules
* Women who were pregnant or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Strumph, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Lexicon Investigational Site, Aurora, Colorado
  - Lexicon Investigational Site, Atlanta, Georgia
  - Lexicon Investigational Site, Baton Rouge, Louisiana
  - Lexicon Investigational Site, Omaha, Nebraska
  - Lexicon Investigational Site, The Bronx, New York
  - Lexicon Investigational Site, Durham, North Carolina
  - Lexicon Investigational Site, Dallas, Texas

REFERENCES:
- [Derived] Sands AT, Zambrowicz BP, Rosenstock J, Lapuerta P, Bode BW, Garg SK, Buse JB, Banks P, Heptulla R, Rendell M, Cefalu WT, Strumph P. Sotagliflozin, a Dual SGLT1 and SGLT2 Inhibitor, as Adjunct Therapy to Insulin in Type 1 Diabetes. Diabetes Care. 2015 Jul;38(7):1181-8. doi: 10.2337/dc14-2806. Epub 2015 Jun 6. PMID 26049551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 sites in United States between 08 February 2013 and 13 January 2014. A total of 36 participants were enrolled and treated in the study which consisted of 2 groups: Pioneer Group and Expansion Groups.
Pre-assignment Details: In this study, first 3 participants (Pioneer Group) received open-label sotagliflozin. Once dosing was completed in Pioneer Group, 33 different participants were randomized in 1:1 ratio to Expansion groups (sotagliflozin or placebo). Randomization was stratified according to baseline glycosylated hemoglobin (A1C [<=8 percent {%} vs. >8%]).
Period: Overall Study
Arm/Group | Sotagliflozin 400 mg - Pioneer Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
Started | 3 | 17 | 16
Completed | 3 | 17 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed using intent-to-treat (ITT) population which consisted of all participants who were randomized in the Expansion Group and participants who received at least 1 dose of study treatment in the Pioneer Group.
Groups:
- Sotagliflozin 400 mg - Pioneer Group: Sotagliflozin 400 mg (two 200 mg tablets), once daily, orally, before breakfast for 29 days; open label administration.
- Total: Total of all reporting groups
Arm/Group | Sotagliflozin 400 mg - Pioneer Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group | Total
Number analyzed (Participants) | 3 | 17 | 16 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (2.08) | 35.6 (11.75) | 38.8 (12.11) | 36.8 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 8 | 19
  Male | 1 | 8 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 2 | 14 | 16 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 172.3 (8.5) | 170.5 (11.7) | 169.5 (12.2) | 170.2 (11.5)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 84.5 (19.2) | 76.8 (15.5) | 78.4 (14.8) | 78.1 (15.1)
Insulin Therapy [Count of Participants; unit: Participants]
  Multiple Daily Injections (MDI) | 0 | 5 | 6 | 11
  Continuous Subcutaneous Insulin Infusion (CSII) | 3 | 12 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Daily Bolus Amount of Exogenous Insulin Required Calculated Over Days 3 to 27 (Treatment Outpatient Period)
Description: Baseline was calculated as the mean value from Day -6 to -2 for Expansion groups and from Day -6 to Day -3 for Pioneer Group. Percent mean change from baseline was calculated as 100*(sum [each daily value - baseline]/number of assessments)/baseline over Days 3 to 27. Least squares (LS) Means and confidence interval (CI) for the Expansion groups were based on an analysis of covariance (ANCOVA) model with covariates of baseline mean total bolus insulin, treatment group, factor used to stratify the randomization (screening A1C <= 8%, > 8%), and random effect of participant*treatment group. LS Means and CI for the Pioneer Group were based on the arithmetic treatment mean.
Time Frame: Baseline, Day 3 to Day 27
Population: Analysis was performed using ITT population. Here, overall number of participants analyzed=participants with available data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sotagliflozin 400 mg - Pioneer Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
Number analyzed (Participants) | 3 | 17 | 15
percent change | -46.32 [-99.71 to 7.06] | -7.00 [-19.18 to 5.17] | -32.14 [-45.09 to -19.18]
Statistical Analysis 1: Comparison: Placebo - Expansion Group vs Sotagliflozin 400 mg - Expansion Group; Between-group comparison of the 2 Expansion Groups was based on an ANCOVA model with covariates of baseline mean total daily bolus insulin, treatment group, factor used to stratify the randomization (screening A1C <= 8%, > 8%), and random effect of participant*treatment group; Test type: Superiority; p = 0.007, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -25.14, 95% CI 2-sided [-42.78 to -7.49] — Difference is sotagliflozin - placebo

2. Secondary Outcome: Percent Mean Change From Baseline in Daily Bolus Amount of Exogenous Insulin Required at Each Meal Calculated Over Days 3 to 27 (Treatment Outpatient Period)
Description: Baseline was calculated as the mean value from Day -6 to -2 for Expansion groups and from Day -6 to Day -3 for Pioneer Group. Percent mean change from baseline was calculated as 100*(sum [each daily value - baseline] / number of assessments)/baseline over Days 3 to 27. Percent change was calculated and is presented separately for each meal: i.e., breakfast, lunch and dinner. LS Means and CI for the Expansion groups were based on an ANCOVA model . LS Means and CI for the Pioneer Group were based on the arithmetic treatment mean.
Time Frame: Baseline, Day 3 to Day 27
Population: Analysis was performed using ITT population. Here, number analyzed=participants with available data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sotagliflozin 400 mg - Pioneer Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
Number analyzed (Participants) | 3 | 17 | 16
percent change
  Before Breakfast: number analyzed (Participants) | 3 | 16 | 14
  Before Breakfast | -42.19 [-169.85 to 85.46] | 10.79 [-13.28 to 34.86] | -25.16 [-51.15 to 0.82]
  Before Lunch: number analyzed (Participants) | 3 | 17 | 15
  Before Lunch | -59.02 [-109.11 to -8.93] | 3.94 [-19.33 to 27.20] | -25.85 [-50.59 to -1.12]
  Before Dinner: number analyzed (Participants) | 3 | 17 | 15
  Before Dinner | -34.83 [-129.08 to 59.42] | 33.34 [-6.53 to 73.22] | -24.02 [-66.57 to 18.54]

3. Secondary Outcome: Percent Change From Baseline in Total Daily Amount of Exogenous Insulin (Total Daily Bolus + Total Daily Basal) Required Calculated Over Days 3 to 27 (Treatment Outpatient Period)
Description: Baseline was calculated as the mean value from Day -6 to -2 for Expansion groups and from Day -6 to Day -3 for Pioneer Group. Percent mean change from baseline was calculated as 100*(sum [each daily value - baseline]/ number of assessments)/baseline over Days 3 to 27. LS Means and CI for the Expansion groups were based on an ANCOVA model. LS Means and CI for the Pioneer Group were based on the arithmetic treatment mean.
Time Frame: Baseline, Day 3 to Day 27
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed=participants with available data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sotagliflozin 400 mg - Pioneer Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
Number analyzed (Participants) | 3 | 17 | 15
percent change | -27.00 [-40.65 to -13.35] | -1.20 [-10.03 to 7.63] | -15.52 [-24.93 to -6.12]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 29
Description: Baseline was defined as the last non-missing assessment prior to first dose of study drug. Change in FPG was calculated by subtracting baseline value from Day 29 value. LS Means and CI for the Expansion groups were based on a linear mixed repeated measures model.
Time Frame: Baseline, Day 29
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligram/deciliter (mg/dL)
Arm/Group | Sotagliflozin 400 mg - Pioneer Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
Number analyzed (Participants) | 3 | 17 | 16
milligram/deciliter (mg/dL) | -54.2 [-85.1 to -23.4] | 10.0 [-9.4 to 29.3] | -12.5 [-36.8 to 11.8]

5. Secondary Outcome: Change From Day 1 in 3-hour Plasma Glucose AUC (AUC0-3 h) Following a Mixed Meal Tolerance Test (MMTT) at Day 29: Expansion Groups
Description: A MMTT with frequent blood sample collection and with urine collection was performed on Day 1 and Day 29. Participants fasted (with the exception of water or non-caffeinated, calorie-free beverages) for at least 8 hours before the start of the MMTT and until the final blood sample was collected. Study drug was to be given within 15 minutes before liquid "Boost® Original" breakfast. The area under the plasma concentration-time curve (AUC) from time-zero to 3h postdose on Day 1 and Day 29 was calculated using the linear-up/log-down trapezoidal rule. Change was calculated by subtracting Day 1 value from Day 29 value. LS Means and CI were based on a linear mixed model.
Time Frame: Prior to start of mixed meal and 30, 60, 90, 120 and 180 min post start of mixed meal, on Day 1 and Day 29
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed=participants with available data for this outcome measure. Data for this outcome measure was not analyzed for Pioneer Group participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg*h/dL
Arm/Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
Number analyzed (Participants) | 16 | 16
mg*h/dL | -140.83 [-225.45 to -56.20] | -308.51 [-393.51 to -223.50]

6. Secondary Outcome: Change From Baseline in Percent Time Per Day Spent in Euglycemic Range (>=70 and <=180 mg/dL) Over Days 3 to 27 (Treatment Outpatient Period) Based on Continuous Glucose Monitoring
Description: Baseline was calculated as the mean value from Day -6 to -2 for Expansion groups and from Day -6 to Day -3 for Pioneer Group. Change in percent time per day spent in euglycemic range was calculated by subtracting baseline value from Day 29 value. LS Means and CI for the Expansion groups were based on a mixed model. LS mean and CI for the Pioneer Group were based on the arithmetic treatment mean.
Time Frame: Baseline, Day 3 to Day 27
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percent time per day
Arm/Group | Sotagliflozin 400 mg - Pioneer Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
Number analyzed (Participants) | 3 | 15 | 13
percent time per day | 6.6 [-31.4 to 44.7] | -1.2 [-6.7 to 4.3] | 11.1 [5.3 to 16.9]

7. Secondary Outcome: Change From Day 1 in 3-hour Urinary Glucose Excretion Following a Mixed Meal Tolerance Test (MMTT) to Day 29: Expansion Groups
Description: A MMTT with frequent blood sample collection and with urine collection was performed on Day 1 and Day 29. Participants fasted (with the exception of water or non-caffeinated, calorie-free beverages) for at least 8 hours before the start of the MMTT and until the final blood sample was collected. Study drug was to be given within 15 minutes before liquid "Boost® Original" breakfast. Participants were asked to void immediately before blood sample 15 minutes before start of mixed meal and immediately after the 180-minute (3 hour) blood sample was collected, and all urine between the -15 minute and post-180-minute time points was collected for urine glucose calculation. Change was calculated by subtracting Day 1 value from Day 29 value. LS Means were based on a linear mixed model.
Time Frame: From 15 minutes before start of mixed meal until 180 min post start of mixed meal, on Day 1 and Day 29
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: gram per 3 hour
Arm/Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
Number analyzed (Participants) | 13 | 16
gram per 3 hour | -6.34 [-20.57 to 7.89] | 8.30 [-4.68 to 21.29]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from Day 1 until the end of study (up to 40 days ).
Description: Safety population included all participants who were randomized and received at least 1 dose of study drug. Participants in this population were assigned to the treatment group as they were treated on Day 1.
Arm/Group | Sotagliflozin 400 mg - Pioneer Group | Placebo - Expansion Group | Sotagliflozin 400 mg - Expansion Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/17 | 2/16
Other Adverse Events (participants affected / at risk) | 1/3 | 12/17 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotagliflozin 400 mg - Pioneer Group (N=3) | Placebo - Expansion Group (N=17) | Sotagliflozin 400 mg - Expansion Group (N=16)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotagliflozin 400 mg - Pioneer Group (N=3) | Placebo - Expansion Group (N=17) | Sotagliflozin 400 mg - Expansion Group (N=16)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ABNORMAL FAECES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FAECES HARD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
LICE INFESTATION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NAIL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NAIL OPERATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 1 (1) | 4 (4)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SINUS HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.